CLINICAL TRIAL: NCT05542225
Title: Effectiveness of Strength Training Versus Flexibility Training in Patients With Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2022/14
Record Dates: First submitted 2022-09-13; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Resistance Training; Standard of Care

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial which will consist of two groups. Once will recieve conventional physcial therapy and the sencond will recieve conventional physcial therapy and slump stretching.Both groups will be recruited concurrently.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be a another person who will be unaware of the group the particpant belong to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional physical therapy with strength training (Experimental): TENS with a frequency of 2-125Hz for about 30mins in prone position. FITT guidelines for strength training: frequency: 2-3 times perweek, time: 3o mins for the whole session, intensity: 8-15 repetitions and type : major muscles( shoulder flexors and extensors, hip and knee flexors, hip abductors and adductors, foot plantar flexors and dorsiflexors using resistance bands)
  Interventions: Procedure: Strength training; Procedure: Standard therapy
- conventional physical therapy with flexibility training (Active Comparator): TENS with a frequency of 2-125 Hz for 30 minutes. FITT guidelines for flexibility; frequency: 5 times per week, intensity: stop before it becomes painful, time: 10-15 minutes,hold for 15 secs and type: major muscle groups( latissmus dorsi, trapezius, gluteus maximus, gluteus medius, gatrocnemius, soleus, hamstringsand paraspinals( errector spinae and multifidus through static stretching technique.
  Interventions: Procedure: Flexibility training; Procedure: Standard therapy

INTERVENTIONS:
Procedure: Strength training — Strength training will be performed with the patient in supine lying position as per FITT guidelines in which resistance will be given with the help of resistance bands on major muscle groups including shoulder flexors and extensors, hip and knee flexors and extensors, hip abductors and adductors,foot plantar flexors and dorsiflexors at an intensity of 8-15 repetitions, 2-3 times per week for 30 minutes.
  Arms: conventional physical therapy with strength training
Procedure: Flexibility training — Flexibility training will be performed with the patient in supine lying position as per FITT guidelines. Static stretching will be applied to the major muscle groups( trapezius, latissmus dorsi, gluteus maximus and medius, gastrocnemus, soleus, hamstrings and paraspinals( errector spinae and multifidi. Session will be completed in 10-15 minutes with a hold of 15 secs, 5 times per week. Stop before it becomes painful.
  Arms: conventional physical therapy with flexibility training
Procedure: Standard therapy — TENS at frequency of 2-125Hz for 30 minutes, pharmacological intervention

SUMMARY:
Fibromyalgia is a rare musculoskeletal condition worldwide.This condition has a significant impact on the person's quality of life by affecting their various activities of daily living. It is a chronic illness characterized by persistent and widespread non-inflammmtory musculoskeletal pain. Various management strategies including both pharmacological and non-pharmacological are used for the treatment of fibromyalgia. In the recent years strength training and flexibility training are being used for the treatment of fibromyalgia. Strength training is used to improve muscle strength, endurance , power or a combination of both, whereas flexibility training is used to improve ability of a joint to maintain the movement. Different studies have shown postive results of strength training and flexibility training in patients with fibromyalgia. However no such study has investigated the combined effects of both theses techniques. So this study aims to investigate the effect of strength training and flexibility training according to the guidelines of FITT protocol.

DETAILED DESCRIPTION:
Fibromyalgia is defined as a chronic illness chracterized by widespread and persistent non-inflammatory musculoskeletal pain including both clinical and emotional symptoms.It is experienced by 2-4.7% of the general population. Commonly it occurs in females as compared to males with a ratio of 3:1 according to ACR criteria 1990.Regarding its clinical features fibromyalgia includes morning stiffness, fatigue, insomnia, mood disorders, anxiety, depression, headaches and other cognitive disorders.Different management strategies including physical therapy are used to treat fibromyalgia. In the recent years strength training and flexibility training are used . strength training is used to improve muscle strength, endurance, power or a combination of both whereas flexibility training improves the mobility of the joint to maintain the movement necessary for carrying out the daily tasks and physical activity. Different studies have shown postive effects of strength training and flexibility training in patients with fibromyalgia. However, there is a lack of literature on the combined effects of strength training and flexibility training according to guidelines of FITT protocol.So this study aims to investigate this aspect.

This Randomized controlled trial will be conducted in Rheumatology Opd of Fauji Foundation hospital using non probability purposive sampling. Initially pilot study with sample size of 10 will be calcullated. Then on the basis of mean difference of participants sample size will be calculated using open epi tool..Patients with diagnosed cases of fibromyalgia in the rheumatology opd of FFH will be recruited according to the eligibility criteria. Participants will be briefed regarding the study objectives, study procedures, risks and benefits of treatment, voluntary participation and right to withdraw. After taking informed consent, basic demographical data and baseline measurements, participants will be randomly allocated into one of the two groups using sealed envelope method. Control group will receive conventional physiotherapy along with flexibility training whereas the experimental group will receive Conventional physiotherapy along with strength training.

Group 1(Control group): TENS at a frequency of 2-125 Hz for 30 minutes, FITT protocol of flexibility training: frequency 5 times per week, intensity: stop before it becomes painful, time: 10-15min, hold for 15 secs and type : major muscle groups( trapezius, latissmus dorsi, gluteus maximus and medius, gastrocnemius, soleus and paraspinals(erector spinae and multifidi) through static stretching.

Group 2(Experimental group): TENS at a frequency of 2-125Hz for 30 minutes, FITT protocol for strength training: frequency 2-3 times per week, intensity :8-15 repetitions, time: 30 minutes for the whole session and type: major muscle groups( shoulder flexors and extensors, hip and knee flexors and extensors,hip abductors and adductors,foot plantar and dorsiflexors using resistance bands.

FREQUENCY:All these measures will be taken at baseline, after two weeks and then after the completion of 4 weeks.

ELIGIBILITY:
Inclusion Criteria

1. Diagnosed cases of fibromyalgia according to diagnostic criteria of ACR 2010 referred from Rheumatology department of FFH.
2. Both males and females adults with an age of 35-60 years

Exclusion Criteria

1. Patients with generalized fatigue
2. Polymyalga rheumatica
3. Hyperthyrodism
4. Regional pain syndrome
5. Irritable bowel syndrome
6. Myofascial pain syndrome
7. Chronic cancer pain
8. Lactating mothers
9. Metabolic disorders

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 4 weeks
  Pain intensity will be measured on numeric rating pain scale. It consists of 11 points( interval 0-10), where 0 corresponds to no pain and 10 corresponds to worst pain imaginable. A graphical representation of 11 spaces is used for patients own evaluation of his or her pain.

SECONDARY OUTCOMES:
Health status | 4 weeks
  Fibromyalgia impact questionnaire (FIQ)
sleep disturbance | 4 weeks
  measured with Medical outcome study sleep scale(MOS)

CONTACTS AND LOCATIONS:
Locations (1):
- Fauji Foundation Hospital, Rawalpindi, Punjab Province, Pakistan